CLINICAL TRIAL: NCT05464238
Title: Implementation, Safety, Tolerability and Effect of Exercise and Respiratory Training on 6-minute Walking Distance in Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction (HFpEF): a Randomized Controlled Multicenter Trial in European Countries.
Brief Title: Training in HFpEF-PH
Acronym: TRAIN HFpEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Head of pulmonary hypertension centre, Thoraxklinik Heidelberg GgmbH, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04ET
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Hypertension Due to Left Heart Disease; Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, parallel-group with crossover of the control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Active Comparator)
  Interventions: Other: Exercise rehabilitation
- Standard treatment (waiting group) (Placebo Comparator)
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Exercise rehabilitation — The initial phase of exercise training will be closely monitored and will be based on a three-weeks in-hospital stay to adjust and teach the exercise training which will be continued at home for 12 more weeks. In-hospital stays will be arranged country specific and hospitalization time may range. The rehabilitation program comprises of interval ergometer training (20 minutes 5 days per week), dumbbell training (30 minutes 5 days per week), respiratory therapy (30 minutes 5 days per week), mental training and guided walks for 2-5 times/week.
  Arms: Exercise training
Other: Standard treatment — Standard treatment during study duration
  Arms: Standard treatment (waiting group)

SUMMARY:
Exercise interventions alone or as a component of a comprehensive cardiac rehabilitation program for patients with heart failure (HFrEF and HFpEF) have already shown to reduce the risk of hospitalisations due to HF and improved exercise capacity and health-related quality of life. Two meta-analyses have confirmed the beneficial effects in cardiorespiratory fitness and quality of life. The effects of exercise training on systolic and diastolic function remain inconclusive. Due to the positive results of exercise training in HFpEF, cardiac rehabilitation is recommended (Class I, level A) to be integrated into the overall provision of HF care. However, none of these studies focused on concomitant PH in HFpEF.

Exercise training in patients with pulmonary hypertension has already shown to improve exercise capacity, quality of life and peak oxygen consumption, which was confirmed by three meta-analyses and a Cochrane review. Though different diagnostic subgroups have already been enrolled in PH exercise training studies, they mainly included pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. Data on combined PH and HFpEF is still lacking.

As recently pointed out by Arena et al. there may thus be an exercise training volume/intensity which may be detrimental to the RV in patients with HF and concomitant PH.

This study is sought to investigate whether a specialized training program is safe and tolerable and may improve exercise capacity, quality of life, hemodynamics, diastolic dysfunction and biomarkers in patients with PH and HFpEF.

DETAILED DESCRIPTION:
During the 6th World Symposium of PH in Nice, three main entities of PH due to left heart disease (PH-LHD) were identified. 1. PH due to HFpEF, 2. PH due to HF with reduced EF (HFrEF) and 3. PH due to valvular disease. The hemodynamic criteria measured by right heart catheterisation (RHC) of PH-LHD include mean pulmonary arterial pressure (mPAP)>20 mmHg and pulmonary arterial wedge pressure (PAWP) >15 mmHg.

The hallmark of HFpEF is an elevation in left-sided filling pressures. In some patients this leads to elevation of mean pulmonary arterial pressure as secondary pulmonary hypertension (PH). Pulmonary arterial pressure is a marker of the severity and chronicity of pulmonary venous congestion in HFpEF and in case of presence of PH, symptoms are more severe and the outcome is poorer.

Recently, an updated diagnostic algorithm (HFA-PEFF) for HFpEF was published as consensus recommendation from the Heart Failure Association of the European Society of Cardiology.

In first step, a pre-test assessment is performed (P: Pretest). In case risk factors for HFpEF are existing electrocardiographic and echocardiographic evaluation as well as an exercise test are required.

If the 1st step is proved positive, a detailed echocardiography (E: echocardiography) should be performed.

A definite diagnosis of HFpEF can be made by right heart catheterization with PAWP ≥15mmHg or LVEDP ≥16mmHg at rest and/or PAWP ≥25mmHg during exercise in presence of preserved left ventricular function.

Exercise interventions alone or as a component of a comprehensive cardiac rehabilitation program for patients with heart failure (HFrEF and HFpEF) have already shown to reduce the risk of hospitalisations due to HF and improved exercise capacity and health-related quality of life . Two meta-analyses have confirmed the beneficial effects in cardiorespiratory fitness and quality of life. The effects of exercise training on systolic and diastolic function remain inconclusive. Due to the positive results of exercise training in HFpEF, cardiac rehabilitation is recommended (Class I, level A) to be integrated into the overall provision of HF care. However, none of these studies focused on concomitant PH in HFpEF.

Exercise training in patients with pulmonary hypertension has already shown to improve exercise capacity, quality of life and peak oxygen consumption, which was confirmed by three meta-analyses and a Cochrane review. Though different diagnostic subgroups have already been enrolled in PH exercise training studies, they mainly included pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. Data on combined PH and HFpEF is still lacking.

In healthy subjects, intensive exercise has already shown to cause potentially deleterious remodeling of the RV. As recently pointed out by Arena et al. there may thus be an exercise training volume/intensity which may be detrimental to the RV in patients with HF and concomitant PH.

This study is sought to investigate whether a specialized training program is safe and tolerable and may improve exercise capacity, quality of life, hemodynamics, diastolic dysfunction and biomarkers in patients with PH and HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥18 years
2. WHO/NYHA functional class II - IV
3. PH with HFpEF diagnosed by right heart catheterisation showing:

   mean pulmonary arterial pressure (mPAP) ≥25mmHg at rest; pulmonary arterial wedge pressure (PAWP) ≥15mmHg at rest or LVEDP ≥16mmHg and/or PAWP≥25 mmHg during exercise, and
4. Preserved left ventricular ejection fraction ≥50%
5. Patients receiving optimized therapy including intensified treatment with diuretics and who have been stable for 1 month before entering the study.
6. Except for diuretics, medical treatment should not be changed during the study period.
7. Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria:

1. Pre-capillary pulmonary hypertension (Group I; Group III; Group IV; Group V according to PH guidelines)
2. Congenital or acquired severe valvular diseases (severe aortic stenosis or insufficiency, severe mitral valve stenosis or insufficiency)
3. Pregnancy or lactation
4. Walking disability
5. Subject who participates in an interventional study during the course of this study
6. Severe lung disease: FEV1/FVC <0.5 and total lung capacity <60% of the normal value
7. Active myocarditis, unstable angina pectoris, exercise induced ventricular arrhythmias, active liver disease, porphyria or elevations of serum transaminases >3 x ULN (upper limit of normal) or bilirubin >1.5 x ULN
8. Haemoglobin concentration less than 75% of the lower limit of normal
9. Systolic blood pressure <85 mmHg
10. History or suspicion of inability to cooperate adequately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance | baseline to 15 weeks

SECONDARY OUTCOMES:
WHO functional class | baseline to 15 weeks
Quality of life physical component scale SF-36 | baseline to 15 weeks
Quality of life mental component scale SF-36 | baseline to 15 weeks
peak oxygen consumption | baseline to 15 weeks
peak oxygen consumption/kg body weight | baseline to 15 weeks
workload achieved during cardiopulmonary exercise testing | baseline to 15 weeks
NT-proBNP (N-terminal pro brain natriuretic peptide) | baseline to 15 weeks
Tricuspid annular plane systolic excursion | baseline to 15 weeks
  echocardiography
Systolic pulmonary arterial pressure | baseline to 15 weeks
  echocardiography
Right atrial area | baseline to 15 weeks
  echocardiography
Right ventricular area | baseline to 15 weeks
  echocardiography
Right ventricular pump function | baseline to 15 weeks
  echocardiography
Left ventricular pump function | baseline to 15 weeks
  echocardiography
Left ventricular eccentricity index | baseline to 15 weeks
  echocardiography

CONTACTS AND LOCATIONS:
Locations (2):
- Centre for Pulmonary Hypertension at the Thoraxklinik Heidelberg, Heidelberg University Hospital, Heidelberg, Germany
- Clinic of Cardiac and Vascular Diseases, Institute of Clinical Medicine, Faculty of Medicine, Vilnius University, Vilnius, Lithuania, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paleviciute E, Celutkiene J, Simbelyte T, Gumbiene L, Jureviciene E, Zakarkaite D, Cesna S, Eichstaedt CA, Benjamin N, Grunig E. Safety and effectiveness of standardized exercise training in patients with pulmonary hypertension associated with heart failure with preserved ejection fraction (TRAIN-HFpEF-PH): study protocol for a randomized controlled multicenter trial. Trials. 2023 Apr 19;24(1):281. doi: 10.1186/s13063-023-07297-x. PMID 37072812